CLINICAL TRIAL: NCT03994237
Title: ALZHEIMER'S CAREGIVER Accompaniment
Brief Title: Accompanying ALZHEIMER CAREGIVER
Acronym: ACCAIDANT
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2016/48
Record Dates: First submitted 2019-05-21; First posted 2019-06-21 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALZHEIMER CAREGIVER: Caregiver available to accompany the patient to the consultation, helping calling for the first time the memory center, aidant who noticed a cognitive disorder help, having a family link identified with the patient
  Interventions: Other: semi-structured interview

INTERVENTIONS:
Other: semi-structured interview — The tool used is a nurse card: there is no validated tool on the expectations of the caregiver in his memory referral. This is a pragmatic and practical questionnaire memory consultation request and domestic life with few items, practical use by telephone.

SUMMARY:
Initiatives have been taken hotline in France and abroad for other conditions, they provide support to patients and their caregivers.

DETAILED DESCRIPTION:
This is a descriptive pilot study, non-interventional, before / after, mono-centric, evaluative, prospective cohort with type score description. The tool used is the grid "mini Zarit", she evaluates the caregiver burden. This grid is enabled in the French version and commonly used in these pathologies.

The evaluation of the quality of life of the caregiver will be performed with the scale "EQ-5D". This tool is easy to use phone, it contains few items. Also there is very little evidence referring to the suffering or negative feelings. It therefore avoids inducing to helping unknown team consultation memory an emotionally negative discourse.

There is no validated tool measuring the service delivered to a nurse hotline. The investigators offer a nurse questionnaire 7 items grouping expectations for the first consultation memory (consultation period, diagnosis, course of the consultation, organization of monitoring). It also provides an update on the daily experiences of the caregiver relative to the organization of care and helped the organization of domestic life of helped.

Nursing questionnaire will assess whether the responses of the nurse in relation to questions about the memory request for consultation were understood in relation to the items. Also, if the caregiver is in support of application in everyday life, the questionnaire will determine if the nursing accompaniment allows the caregiver to acquire knowledge or skills, or better organization of everyday life. The question of the entourage of the caregiver assesses the isolation level of the caregiver and whether the environment is not mobilized or after an update with the nurse.

If help is hospitalized, the pattern will be recovered. The Scientific Council will assess whether the information collected and the information provided would have prevented it.

ELIGIBILITY:
Inclusion Criteria:

* Helping with age ≥ 18 years
* Helping speak and understand the French
* Help available to accompany the patient to the consultation
* Helping calling for the first time the memory center
* Helping who noticed a cognitive disorder in assisted
* Age over 75 years
* beneficiary or affiliated to a social security scheme Patient
* Patient with a cognitive disorder noticed by the caregiver

Exclusion Criteria:

* Helping placed under judicial protection
* Any medical or paramedical personnel in connection with the care of a nursing home eligible patient (Accommodation Establishment for dependent elderly, hospital, SSR (Care and Rehabilitation Services), institutional caregivers,
* private health professionals, such as neighborhood (doctor, nurse liberal, physiotherapist
* Neighborhood.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Helping with age ≥ 18 years, speaking and understanding the French and available to accompany the patient to the consultation
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
score of the grid "MiniZarit" | Month 1
  The evaluation of the quality of life of the caregiver, score between 0 and 7. point for positive response for difficulties in family life, difficulties in relationships with friends, hobbies, or in your job, a repercussion on health (physical and / or psychological), feeling that caregiver is no longer recognizing his parent, he afraid for the future of his parent, he would like to be (more) helped to take care of his parent, he feel a burden in taking care of his parent.
score of the EuroQuol scale | Month 1
  The evaluation of the quality of life of the caregiver
  The point repartition :
  Mobility (1 point : to have no problem getting around on foot ; 2 : to have problems getting around on foot; 3. to oblige to remain in bed) Self-sufficiency (1 point : to have no problem taking care of myself; 2 : to have problems washing or dressing myself alone;3 : to be unable to wash or dress myself alone) Regular activities (1 point : to have no problem performing my daily activities (eg work, study, housework, family activities or hobbies) ;2. : to have problems to perform my day-to-day activities;3. : to be unable to perform my normal activities.) Pain / discomfort (1. : to have no pain or discomfort; 2. : to have moderate pain or discomfort (s), 3. : to have severe pain or discomfort (s)) Anxiety / Depression (1. : to be not anxious or depressed; 2. : to be moderately anxious or depressed ;3. : to be extremely anxious or depressed)

SECONDARY OUTCOMES:
Number of days between pre-clinical consultation and consultation MEMORY | Month 3
  Impact of pre-clinical consultation on information support in consultation MEMORY
Questionnary for caregivers' organization | Day 1
  Evalution of professional helpers, number of technical assistance (remote alarm ...), nature of handicap , presence of correction device, number of taking medication drugs, Sleep is good or not, recent weight evolution
Questionnary for caregivers' organization | Month 1
  Evalution of professional helpers, number of technical assistance (remote alarm ...), nature of handicap , presence of correction device, number of taking medication drugs, Sleep is good or not, recent weight evolution

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle GUILLARD, Principal Investigator — University of Bordeaux
Locations (1):
- CHU de Bordeaux, Pessac, France